CLINICAL TRIAL: NCT07342010
Title: Evaluation of the Effect of Lidocaine With Adrenaline, With or Without Bicarbonate, on Early Postoperative Recovery in WALLANT-type Outpatient Hand and Foot Surgery: A Prospective, Randomised, Double-blind, Single-centre Non-inferiority Study.
Brief Title: Bicarbonate Addition to Lidocaine-Epinephrine in Surgery Under WALANT
Acronym: ROPIWA-2
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-519650-36-00
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia, Local; Hand Surgery; Foot Surgery; Walant Surgery
Keywords: lidocaine,; bicarbonates,; Quality of recovery; Walant
MeSH Terms: interventions — Epinephrine; Bicarbonates

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, randomized (1:1 ratio), double-blind, noninferiority trial comparing two WALANT solutions (with or without bicarbonate addition) in patients scheduled for distal hand or foot ambulatory surgery.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to the WALANT local infiltration solution administered.
  Investigators performing the local anesthesia and the surgical procedure, as well as outcome assessors (investigator-delegated evaluators, hospital clinical research associates, and evaluating physicians), will also be blinded to treatment allocation. Preoperative and postoperative assessments will be performed by providers different from those who performed the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients undergoing hand and foot surgery with lidocaine and Epinephrine alone (Experimental): Patients undergoing hand and foot surgery under WALANT using lidocaine 5 mg/mL combined with epinephrine 0.005 mg/mL, without bicarbonate.
  Interventions: Combination Product: Ambulatory surgery under Lidocaine with epinephrine alone
- Patients undergoing hand and foot surgery with buffered lidocaine (Active Comparator): Patients undergoing hand and foot surgery under WALANT using lidocaine 5 mg/mL combined with epinephrine 0.005 mg/mL, with bicarbonate.
  Interventions: Combination Product: Ambulatory surgery under lidocaine with epinephrine plus bicarbonate

INTERVENTIONS:
Combination Product: Ambulatory surgery under Lidocaine with epinephrine alone — The anesthetic solution will consist of lidocaine 5 mg/mL combined with epinephrine 0.005 mg/mL, administered as 18 mL (90 mg of lidocaine) plus 2 mL of saline (placebo), for a total volume of 20 mL Additional solution will be administered if sensory block is insufficient prior to incision.
  Other Names: Local infiltration with lidocaine-epinephrine
  Arms: Patients undergoing hand and foot surgery with lidocaine and Epinephrine alone
Combination Product: Ambulatory surgery under lidocaine with epinephrine plus bicarbonate — The anesthetic solution will consist of lidocaine 5 mg/mL combined with epinephrine 0.005 mg/mL, administered as 18 mL (90 mg of lidocaine) plus 2 mL of 8.4% bicarbonate, for a total volume of 20 mL.
  Additional solution will be administered if sensory block is insufficient prior to incision.
  Other Names: Local infiltration with lidocaine-epinephrine and bicarbonate
  Arms: Patients undergoing hand and foot surgery with buffered lidocaine

SUMMARY:
Distal upper limb and distal lower limb surgery performed under local anesthesia using the WALANT technique (Wide Awake Local Anesthesia No Tourniquet) has become standard practice in ambulatory orthopedic surgery. Current infiltration mixtures used by orthopedic surgeons include lidocaine-epinephrine with the addition of 8.4% bicarbonate to reduce injection-related pain and improve analgesia duration. However, the clinical benefit of bicarbonate addition remains insufficiently supported by evidence and may increase preparation complexity and risk, including potential solution crystallization.

The aim of the ROPIWA-2 trial is to investigate whether omission of bicarbonate from the local infiltration mixture is noninferior to bicarbonate addition with respect to early postoperative quality of recovery on postoperative day 1. We hypothesize that removing bicarbonate does not impair postoperative quality of recovery after ambulatory hand and foot surgery under WALANT. Expected benefits include confirmation of a simpler, ready-to-use anesthetic solution that is easier and safer to use, without reducing patient comfort or recovery. The expected risks are those normally associated with this type of procedure.

DETAILED DESCRIPTION:
Study context WALANT (Wide Awake Local Anesthesia No Tourniquet) is increasingly used for ambulatory hand and foot surgery, as it allows surgery without preoperative fasting and provides effective local anesthesia without a tourniquet, while promoting early functional recovery.

Sodium bicarbonate is commonly added to lidocaine-epinephrine solutions to reduce injection-related pain and prolong the duration of the anesthetic block. However, its clinical benefit remains uncertain and may increase preparation complexity.

Therefore, a robust methodological assessment of the impact of bicarbonate omission on early postoperative recovery is warranted in ambulatory WALANT surgery.

Primary objective To evaluate the effect of two WALANT local anesthesia protocols (lidocaine-epinephrine with or without bicarbonate addition) on early postoperative recovery at 24 hours after ambulatory hand and foot surgery.

Key secondary objectives A) Sensory block onset time. B) Intraoperative anesthetic block failure rate. C) Pain related to injection of the WALANT anesthetic solution. D) Intraoperative pain intensity. E) Patient satisfaction with perioperative care. F) Postoperative pain scores. G) Postoperative analgesic consumption, including opioids. H) Duration of the anesthetic block I) Postoperative adverse events.

Study design and conduct This prospective, single-center, randomized, double-blind, noninferiority trial will compare two 20 mL WALANT (Wide Awake Local Anesthesia No Tourniquet) solutions in patients scheduled for distal hand or foot ambulatory surgery.

The intervention group will receive lidocaine 5 mg/mL combined with epinephrine 0.005 mg/mL (18 mL of solution mixed with 2 mL of saline as placebo), whereas the control group will receive a similar solution including 8.4% bicarbonate (18 mL of solution mixed with 2 mL of bicarbonate). Both solutions will be administered by orthopedic surgeons prior to surgical incision.

Additional solution will be administered if sensory block is insufficient prior to incision.The maximum total lidocaine dose per patient will not exceed 800 mg in adults, in accordance with the approved labeling and standard clinical use of the drug.

Adults (≥18 years) eligible for ambulatory WALANT procedures (hand or selected foot surgeries) will be screened during the preoperative orthopedic consultation (pre-inclusion visit). All eligible patients will receive oral and written information, with at least one day between the pre-inclusion and inclusion visits to allow time for reflection and informed consent.

After written consent is obtained, patients will be randomized in a 1:1 ratio to the control group (with bicarbonate) or the intervention group (without bicarbonate). The surgical procedure under WALANT will be performed by orthopedic surgeon investigators.

Preoperative pain intensity (NRS), surgery-related anxiety (NRS), and the QuickDASH score will be recorded prior to the surgical procedure. Before hospital discharge, postoperative pain and patient satisfaction will be assessed. All patients will receive a standardized postoperative analgesic regimen.

Postoperative follow-up calls conducted by the clinical research associate will occur at 24 hours (NRS pain score, QoR-15 score, duration of the analgesic block, analgesic consumption, and adverse events) and at 48 hours (NRS pain score and adverse events). Study participation will end after the 48-hour follow-up call.

The estimated sample size is 150 patients, with 75 patients in each study arm. For the primary outcome, the noninferiority margin for the QoR-15 score is set at 6 points.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) eligible for ambulatory surgery under WALANT for Hand surgery (including carpal tunnel release, trigger finger release, or Dupuytren's disease surgery) and foot surgery (including hallux valgus or hallux rigidus.)
* Provision of free and informed consent.
* Signed informed consent form.
* Affiliation with or beneficiary of a health insurance system

Exclusion Criteria:

* Ischemic vascular disorders, including severe Raynaud's disease, Buerger's disease, or diabetic microangiopathy.
* Scleroderma.
* Known allergy to lidocaine or potential cross-reactivity with other amide-type local anesthetics.
* Severe hepatic impairment.
* Acute porphyria.
* Intravascular administration of local anesthesia.
* Local anesthetic infiltration at the level of the extremities.
* Coronary artery disease.
* Ventricular arrhythmias.
* Severe arterial hypertension.
* Obstructive cardiomyopathy.
* Hyperthyroidism.
* Hypovolemia.
* Participation in an interventional clinical research study classified as category 1 (RIPH category 1).
* Ongoing exclusion period related to participation in another clinical study.
* Legal protection status (guardianship, trusteeship, or judicial protection).
* Inability to provide informed consent.
* Inability to receive or understand adequate study information.
* Pregnancy, labor, or breastfeeding. Women of childbearing potential will undergo a urine pregnancy test prior to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
QoR-15 score, assessed at 24 hours postoperatively in both study arms | 24 hours after surgery
  QoR-15 score, assessed at 24 hours postoperatively in both study arms. This validated questionnaire includes 15 items covering five dimensions: pain, physical comfort, physical independence, psychological support, and emotional state. Each item is rated on a 1-10 scale, with a total score ranging from 15 to 150.

SECONDARY OUTCOMES:
Sensory block onset time | Day 0
  Anesthetic block onset time: time (in minutes) from the initial injection to complete sensory block of the surgical area, defined as absence of sensation to pinprick testing performed at 5-minute intervals by the surgeon.
Intraoperative anesthetic block failure rate | Day0
  Defined as the need for rescue intraoperative reinjection of local anesthetic solution by the surgeon due to persistent sensation during anesthetic block testing using nociceptive stimuli (yes/no).
Pain related to injection of the WALANT anesthetic solution. | Day 0
  Patient self-assessment of pain experienced during WALANT administration, measured using a Numeric Rating Scale (NRS) from 0 (no pain) to 10 (worst imaginable pain).
Intraoperative pain intensity | Day 0
  Patient self-assessment of pain experienced during the surgical procedure, measured using a Numeric Rating Scale (NRS) from 0 (no pain) to 10 (worst imaginable pain).
Patient satisfaction with perioperative care | Day 0
  Patient self-assessment of satisfaction with perioperative management, measured using a Numeric Rating Scale (NRS) from 0 (not satisfied at all) to 10 (completely satisfied).
Postoperative pain scores | Day 2
  Patient self-assessment of pain intensity measured using a Numeric Rating Scale (NRS) from 0 (no pain) to 10 (worst imaginable pain) at postoperative day 0 (hospital discharge), postoperative day 1, and postoperative day 2.
Postoperative analgesic consumption, including opioids | Day 2
  Total consumption (in milligrams) of paracetamol and ketoprofen during the first 48 postoperative hours, as well as tramadol consumption (in milligrams) during the same period.
Duration of the anesthetic block | Day 1
  Time (in minutes) from the initial anesthetic solution injection to block resolution, defined by the patient-reported onset of postoperative pain (patient self-assessment).
Postoperative adverse events | Day 2
  Occurrence (yes/no) of the following postoperative complications from surgery to postoperative day 2:: hematoma, bleeding, wound dehiscence, paresthesias, nausea, vomiting, rehospitalization, surgical site infection, or other postoperative complications.

OTHER OUTCOMES:
Sex of patients | Day 0
  Male/Female
Age of patients | Day 0
  In years
Weight of patients | Day 0
  In kilograms
Height of patients | Day 0
  In centimeters
Type of surgery | Day 0
  Description of the surgery.
Current medications | Day 0
  Current medications, including anticoagulants and preoperative pain medications.
Medical history | Day 0
  Medical history, including smoking status, diabetes mellitus, arterial hypertension, peripheral arterial disease, and peripheral neuropathy.
QuickDASH score (if hand surgery) | Day 0
  QuickDASH (short version of DASH - Disabilities of the Arm, Shoulder and Hand) is a self-assessment questionnaire designed to measure functional limitations and symptoms related to musculoskeletal disorders of the upper limb.
Socioprofessional category | Day 0
  Socioprofessional category recorded according to predefined categories (employed, unemployed, retired, or student).
Preoperative surgery-related anxiety | Day 0
  Patient self-assessment measured using a Numeric Rating Scale (NRS) from 0 (no anxiety) to 10 (maximum anxiety) prior to surgery
Preoperative pain related to the surgical indication | Day 0
  Preoperative pain related to the surgical indication: measured using a Numeric Rating Scale (NRS).
Chronic pain related to the surgical condition | Day 0
  Presence of pain lasting more than 3 months prior to surgery
Surgical laterality | Day 0
  Surgical laterality: right or left side and Handedness: right-handed or left-handed

CONTACTS AND LOCATIONS:
Locations (1):
- Yann GRICOURT, Nîmes, Gard, France

IPD SHARING:
Plan to Share IPD: Undecided